CLINICAL TRIAL: NCT07204223
Title: Comparison of the Tulip Airway and the Guedel Airway in Anticipated Difficult Mask Ventilation: A Prospective, Randomized, Controlled Crossover Trial
Brief Title: Tulip Airway in Difficult Mask Ventilation (TADMV)
Acronym: TADMV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ayse Zeynep Turan Civraz (Other Government)
Responsible Party: Sponsor-Investigator, Ayse Zeynep Turan Civraz, Assoc.Prof., Kocaeli City Hospital
Organization: Kocaeli City Hospital (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: KSH- AZTC- 02
Record Dates: First submitted 2025-09-11; First posted 2025-10-02 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Difficult Mask Ventilation; Airway Devices
Keywords: guedel airway; airway management; difficult bag mask ventilation; tulip airway

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guedel Group (Active Comparator): Guedel airway will be the first device during mask ventilation
  Interventions: Device: Guedel Airway
- Tulip Group (Experimental): Tulip airway wil be the initial device for mask ventilation
  Interventions: Device: Tulip Airway

INTERVENTIONS:
Device: Tulip Airway — In this study, patients scheduled for surgery under general anesthesia who meet the criteria for anticipated difficult mask ventilation will be included. Randomization will be performed to determine which device will be used first. If the Tulip airway is selected as the first device in the randomization process, mask ventilation will be initiated with the Tulip airway.
  Arms: Tulip Group
Device: Guedel Airway — In this study, patients scheduled for surgery under general anesthesia who meet the criteria for anticipated difficult mask ventilation will be included. Randomization will be performed to determine which device will be used first. If the Guedel airway is selected as the first device in the randomization process, mask ventilation will be initiated with the Guedel airway.
  Arms: Guedel Group

SUMMARY:
During surgery, right after anesthesia is given, the first step to help the patient breathe is to provide breathing support with a mask. This step is very important because if there is a problem with mask ventilation, the anesthesia team must quickly use other methods to help the patient breathe.

For some people, mask ventilation can be more difficult. Factors such as older age, having a beard, missing teeth, being overweight, sleep apnea, or certain facial shapes can make this process harder.

To make mask ventilation easier, special devices placed in the mouth are used. The most common one is called the Guedel airway. In recent years, a new device called the Tulip airway has also been introduced. The shape and features of the Tulip airway are designed to make breathing support easier.

In this study, we will compare the Tulip airway and the Guedel airway in patients who are expected to have more difficult mask ventilation. Our goal is to find out which device makes it easier and safer to help patients breathe.

DETAILED DESCRIPTION:
The first step in airway management following anesthesia induction is the period of bag-mask ventilation. This step is the most critical phase of airway management because, if mask ventilation fails, the anesthesiologist must make a life-saving decision for the patient. Bag-mask ventilation is a technical skill acquired over time; therefore, difficulty in mask ventilation may be related to either the provider or the patient. According to the literature, the incidence of difficult mask ventilation varies between 0.08% and 15% in different studies.

The American Society of Anesthesiologists (ASA) defines difficult mask ventilation as inadequate mask or supraglottic airway (SGA) ventilation, excessive air leakage, or excessive resistance to airflow during inspiration or expiration. Signs of inadequate ventilation include, but are not limited to, absent or insufficient chest movement, absent or diminished breath sounds, auscultatory signs of severe obstruction, cyanosis, gastric insufflation or distension, decreased or inadequate oxygen saturation (SpO₂), absence or inadequacy of end-tidal carbon dioxide (EtCO₂), absence or inadequacy of expiratory gas flow on spirometry, and hemodynamic changes associated with hypoxemia or hypercarbia (e.g., hypertension, tachycardia, arrhythmia).

Predictors of difficult mask ventilation include age over 55 years, the presence of a beard, poor mask fit due to secretions, edentulism, a history of snoring or obstructive sleep apnea syndrome (OSAS), and obesity. In anesthesia practice, when faced with difficult mask ventilation, various maneuvers, two-hand techniques, and adjunct airway devices are employed. Among these devices are various oral airways, the most common of which is the Guedel airway.

In recent years, new oral airway devices have been introduced as alternatives to the Guedel airway. The Tulip airway is a novel oral airway that is longer than the Guedel airway, equipped with a cuff, and features a connector that allows attachment to the breathing circuit. These characteristics enable it to be secured within the oral cavity via its cuff, and connection to the breathing circuit allows for airway management that may be more comfortable for the anesthesiologist compared to two-handed mask control.

The superiority of the Tulip airway over the Guedel airway has been demonstrated in patients with cervical spine injury, in edentulous manikins, and in patients undergoing general anesthesia. However, it has not been studied in patients with anticipated difficult mask ventilation. The aim of our study is to investigate whether the Tulip airway provides superior performance to the classical Guedel airway during the mask ventilation phase in patients with anticipated difficult mask ventilation. We hypothesize that the use of the Tulip airway in such patients will improve respiratory parameters and reduce the risk of complications during mask ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years
* Patients scheduled for elective surgery under general anesthesia
* Patients with at least two risk factors for difficult mask ventilation, including:
* Age over 55 years
* Presence of beard
* Edentulism (missing teeth)
* Obesity (Body Mass Index (BMI) ≥ 30 kg/m²)
* History of obstructive sleep apnea syndrome (OSAS) or snoring
* Neck circumference > 43 cm
* Retrognathia (small jaw structure)
* Patients classified as American Society of Anesthesiologist (ASA) physical status 1, 2, or 3
* Patients who provide informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients with a history of airway surgery (e.g., tracheostomy, maxillofacial surgery)
* Patients with severe cardiopulmonary diseases (e.g., advanced Chronic obstructive Pulmonary Disease (COPD), pulmonary hypertension, severe heart failure)
* Patients with craniofacial anomalies or significant anatomical airway deformities
* Patients requiring emergency surgery
* Patients with gastroesophageal reflux disease (GERD) and high risk of aspiration
* Patients with active upper respiratory tract infection
* Patients with a history of difficult intubation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Expiratory Tidal Volume | Minute 5
  Patients in Group G will have a Guedel airway placed in a size appropriate for their weight, and the practitioner will hold the mask with both hands. Patients in Group T will have a Tulip airway placed in a size appropriate for their weight. In both groups, to prevent variability on the part of the practitioner, patients will be ventilated in pressure-controlled mode at 15 (centimeters of water) cmH₂O pressure, respiratory rate 10 breaths/min, an I:E ratio of 1:3, and an oxygen flow rate of 10 L/min without Positive End Expiratory Pressure (PEEP). For both groups, successful mask ventilation will be defined as a tidal volume (TV) of at least 250 ml.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Z Turan Cıvraz, Assoc. Prof., Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) underlying the findings of this study will be available upon reasonable request from qualified researchers, after de-identification, beginning 6 months following publication and ending 5 years later. Data will be shared for academic purposes with appropriate ethical approval and a signed data access agreement."

REFERENCES:
- [Background] Shaikh A, Robinson PN, Hasan M. The Tulip GT(R) airway versus the facemask and Guedel airway: a randomised, controlled, cross-over study by Basic Life Support-trained airway providers in anaesthetised patients. Anaesthesia. 2016 Mar;71(3):315-9. doi: 10.1111/anae.13328. Epub 2015 Dec 19. PMID 26684684
- [Background] Imashuku Y, Kitagawa H, Mizuno T. Usefulness of Tulip Airway in Edentulous Elderly Patients. Anesth Prog. 2022 Sep 1;69(3):9-12. doi: 10.2344/anpr-69-01-01. PMID 36223186
- [Background] Koga K, Sata T, Kaku M, Takamoto K, Shigematsu A. Comparison of no airway device, the Guedel-type airway and the Cuffed Oropharyngeal Airway with mask ventilation during manual in-line stabilization. J Clin Anesth. 2001 Feb;13(1):6-10. doi: 10.1016/s0952-8180(00)00228-2. PMID 11259887
- [Background] Apfelbaum JL, Hagberg CA, Caplan RA, Blitt CD, Connis RT, Nickinovich DG, Hagberg CA, Caplan RA, Benumof JL, Berry FA, Blitt CD, Bode RH, Cheney FW, Connis RT, Guidry OF, Nickinovich DG, Ovassapian A; American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Practice guidelines for management of the difficult airway: an updated report by the American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Anesthesiology. 2013 Feb;118(2):251-70. doi: 10.1097/ALN.0b013e31827773b2. No abstract available. PMID 23364566
- [Background] Bradley P, Chapman G, Crooke B, Greenland K. Airway Assessment.
- [Background] Bucher JT, Vashisht R, Cooper JS. Bag-Valve-Mask Ventilation. 2025 May 3. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK441924/ PMID 28722953